CLINICAL TRIAL: NCT04765930
Title: Combined Q-switched Nd:YAG Laser and Platelet Rich Plasma Versus Q- Switched Nd:YAG Laser Alone in the Treatment of Melasma: A Split Face Study.
Brief Title: Combined Q-switched Nd:YAG Laser and Platelet Rich Plasma Versus Q- Switched Nd:YAG Laser Alone in Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona El-Kalioby, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MelaPRP2020
Record Dates: First submitted 2021-02-04; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Hyperpigmentation; Melasma; PRP; Lasers
Keywords: laser toning; Hemi-MASI; Colorimeter; Erythema Index; Melanin Index
MeSH Terms: conditions — Hyperpigmentation; Melanosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Injection (Active Comparator): Half of the face
  Interventions: Other: Q-switched nd:YAG laser toning
- Saline injection (Placebo Comparator): Other half of the face
  Interventions: Other: Q-switched nd:YAG laser toning

INTERVENTIONS:
Other: Q-switched nd:YAG laser toning — Q-switched nd:YAG laser toning for melasma.

SUMMARY:
Melasma is a common, acquired, esthetically disfiguring hypermelanosis of the face. Melasma is considered a disappointing challenge when treatment options are addressed. Diverse treatment modalities such as retinoic acid, hypo-pigmenting agents like hydroquinone, azelaic acid, and kojic acid, chemical peels, microdermabrasion, and lasers have been tried for the treatment of melasma. There is no universally proven therapy that induces and maintains remission of the condition. Q-switched: Nd YAG laser toning and platelet rich plasma (PRP) are promising treatments for melasma.The aim of this work is evaluate the efficacy and safety of combined PRP and Q-switched: NdYAG laser in the treatment of melasma using clinical assessment, in addition to assessment of Melanin Index and Erythema Index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral nearly symmetric melasma on the face.

Exclusion Criteria:

* Patients receiving systemic or topical or laser treatment relevant to melasma within three months before enrollment into the study.
* Use of oral or injectable contraceptives or hormone replacement therapy during treatment or 12 months before
* Patients active skin infections and active HSV
* History of hypertrophic scars or keloids.
* Patients with hypercoagulable state or bleeding diatheses
* Pregnant and lactating females.
* History of liver diseases
* Intake of systemic chemotherapy, corticosteroids, antiplatelets or anticoagulants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemi-Melasma Area and Severity Index (MASI) score | 2 months after final treatment
  Hemi-Melasma Area and Severity Index(MASI) score for Pigmentation, and Area of involvement. The minimum value is 0 and the maximum value is 12. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Melanin Index | 2 months after final treatment
  Objective assessment of melanin index using colorimeter apparatus. The minimum value is 0. No maximum value. Higher scores mean a worse outcome.
Erythema Index | 2 months after final treatment
  Objective assessment of erythema index using colorimeter apparatus. The minimum value is 0. No maximum value. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Paients' Satisfaction assessed by the VAS | 2 months after final treatment
  a four-scale grading score: poor: response rate= 0-25%; fair: response rate= 25-50%; good: response rate=50-75%; excellent: response rate=75-100%

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes